CLINICAL TRIAL: NCT00860691
Title: Double Blinded Randomized Clinical Trial of the Effect of Open Versus Laparoscopic Colectomy on Neutrophils in Patients With Colon Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Dubrava (Other)
Collaborators: Ministry of Science, Education and Sport, Republic of Croatia (Other Government)
Responsible Party: Professor Igor Stipancic, MD, PhD, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 198-0000000-3104
Record Dates: First submitted 2009-03-10; First posted 2009-03-12 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2010-03

CONDITIONS: Colonic Neoplasms
Keywords: Curative surgical resection; Laparoscopic technique
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ARM I - Open colorectal surgery (Active Comparator): Open colorectal surgery
  Interventions: Procedure: Therapeutic conventional colorectal surgery
- ARM II - Laparoscopic colorectal surgery (Experimental): Laparoscopic colorectal surgery
  Interventions: Procedure: Therapeutic laparoscopic colorectal surgery
- Control - reference value (Other): Blood samples from healthy volunteers will be obtained at one time point.Peripheral blood samples will be obtained into tubes with no additive (BD Vacutainer System, Plymouth, UK).Samples will be processed to serum. Serum concentrations of sFas will be quantitative determinated by a sandwich enzyme immunoassay technique (ELISA)using specific anti-Fas MoAbs, Human sFas Immunoassay. Serum concentrations of sFasL will be quantitative determinated by a sandwich enzyme immunoassay technique (ELISA) using specific anti-Fasl MoAbs, Human sFas Immunoassay. Serum concentration of IL - 17 will be quantitative determinated by a sandwich enzyme immunoassay technique (ELISA) using Human IL-17 Immunoassay. . Peripheral blood samples for measurement of oxidative burst in neutrophils will be collected into heparinised blood tube. burst neutrophil production will be determined quantitatively by flow cytometry as described by Rothe using a commercial kit Bursttest Kit.
  Interventions: Other: Peripheral blood sampling and performing: ELISA test of sFas, sFasL, IL - 17 and Bursttest

INTERVENTIONS:
Procedure: Therapeutic conventional colorectal surgery — Patients with colorectal cancer undergo open laparotomy and colorectal resection
  Other Names: Open colorectal surgery
  Arms: ARM I - Open colorectal surgery
Procedure: Therapeutic laparoscopic colorectal surgery — Patients with colorectal cancer undergo laparoscopic colorectal resection
  Arms: ARM II - Laparoscopic colorectal surgery
Other: Peripheral blood sampling and performing: ELISA test of sFas, sFasL, IL - 17 and Bursttest — Informed consent will be obtained.Blood samples will be obtained at one time point. .Samples will be processed to serum, using a refrigerated centrifuge, then stored at -80C until analysis. Peripheral blood samples for measurement of oxidative burst in neutrophils will be collected into heparinised blood tube.Serum concentrations of sFas will be quantitative determinated by a sandwich enzyme immunoassay technique (ELISA) using specific anti-Fas MoAbs, Human sFas Immunoassay (Code: DFS00; QUANTIKINE R&D Systems Inc, Minneapolis, USA). Serum concentrations of sFasL will be quantitative determinated by a sandwich enzyme immunoassay technique (ELISA) using specific anti-Fasl MoAbs, Human sFas Immunoassay (Code: DFS00; QUANTIKINE R&D Systems Inc, Minneapolis, USA).Respiratory burst neutrophil production will be determined quantitatively by flow cytometry using a commercial kit Bursttest Kit (Cat. No: 10-0200; ORPEGEN Pharma, Germany)
  Arms: Control - reference value

SUMMARY:
The purpose of this study is:

* to determine neutrophil activity in patients with colon cancer,
* to determine levels sFas, sFasL and IL - 17 in serum of healthy volunteers and colon cancer patients and establish its prognostic value,
* to elucidate the relationship between serum sFas, sFasL and IL - 17 levels and clinicopathologic features of colon cancer,
* to compare the influence of laparoscopic and conventional procedures on postoperative serum sFas and sFasL levels in colon cancer patients
* to compare the influence of laparoscopic and conventional procedures on postoperative serum IL - 17 levels in colon cancer patients
* to compare the influence of laparoscopic and conventional procedures on postoperative neutrophil functions
* to confirm the expression of FasL protein in human colorectal cancer and elucidate the relationship between FasL expression and clinicopathologic features of the disease, to establish the prevalence of Fas in primary colon adenocarcinomas and elucidate the relationship between FasL expression and clinicopathologic features of the disease
* to determine the functional activity of tumour infiltrating neutrophils

DETAILED DESCRIPTION:
Colorectal cancer is the leading cause of death worldwide. Tumour cell extravasation plays a key role in tumour metastasis. There are evidences tumour cell-leukocyte interactions may support tumour cell invasion and could create an optimal microenvironment for tumour growth at the metastatic site. Neutrophils produce free radicals and proteases; they could cause tumour cytolysis, as well as promote tumour growth and metastasis. It seems that neutrophils play an important role in the context of tumour and angiogenesis.

It is not well understood why FasL induces immune privilege in some organs but elicits inflammation. To explain these apparently conflicting phenomena, it is important to investigate the mechanism of FasL-induced inflammation in detail. Fas/FasL can serve as potential targets for effective antitumor therapy. This research will be useful to eludicate the importance of neutrophil in colorectal cancer. We will investigate the possible role of neutrophil activity and FasL-induced neutrophil infiltration on tumor growth in colorectal cancer. sFas and sFasL could be a way to measure the balance of apoptotic and immunoescape effect after surgical resection of colon cancer.

If the number of neutrophils in peripheral blood mirrors the situation in the tumor tissue, these data could support the investigation of neutrophil-targeted therapies in anti-cancer strategy.

Inflammation-dependent angiogenesis seems to be a central force in tumor growth and expansion, a concept supported by the observation that the use of anti-inflammatory drugs, leads to angiogenesis inhibition. The mechanisms of inflammatory angiogenesis could provide new approaches to target, cure, or prevent tumor angiogenesis. Investigation of the physiologic regulation of IL-17 may thus be useful for the treatment in clinical settings characterized by persistent neovascularisation.

Inhibition of neutrophil elastase might not only reduce the inflammatory response, but could also prevent cancer cell progression. Anti-neutrophil elastase therapy after tumour resection might be an important strategic approach for managing postoperative complications and preventing cancer recurrence.

Patients will be allocated to laparoscopic or conventional open colorectal surgery after eligibility had been confirmed and informed consent given. Randomization will be performed by computer; sequencing was based on a list of variable block sizes for a single centre without further stratification. The randomization list and opaque envelopes will be generated by independent personnel not otherwise involved in the trial. Information on the operation will be remain in consecutively numbered and sealed envelopes that will be stored in a specific box at the clinical site. The envelope containing the allocation will be added to a patient's file shortly before he or she enter the operating theatre. The envelope will be then open and the surgeon will perform the assigned procedure. Until the day of discharge of participants, nurses and other medical staff will be blinded for the type of surgery performed in patients with colorectal cancer by applying a covering abdominal bandage.

During the trial, all blood samples will be retrieved and assessed by a cytologist and molecular biologist blinded to the study arms.

ELIGIBILITY:
Inclusion Criteria:

All patients will be informed that additional blood and tissue samples will be taken during perioperative period for colon cancer research, and written consent will be obtained. Informed consent will be also obtained from each healthy volunteer.

Patients with the clinical diagnosis of colorectal cancer based on colonoscopy following histological confirmation will recruited. They should be suitable for elective surgical resection of the tumour along with lymph node dissection by right and left hemicolectomy, sigmoid colectomy, and anterior resection. Clinicopathologic characteristics of these patients will be investigated based on TNM classification of malignant tumours and modified Dukes classification Inclusion criteria; age between 18 and 80 years; colorectal cancer with single tumour locating at cecum, ascending colon, descending colon, sigmoid colon or recto sigmoid junction (distance from anal verge more than 15 cm); ASA I-III; and informed consent.

Exclusion criteria; patient refusal to participate in the prospective data collection; prior midline laparotomy; emergency surgery or urgent operation within 24 h after admission to the hospital; conversion to laparotomy; mechanic ileus; perforation or abscess with septic inflammatory response syndrome; planned stoma, low anterior resection or rectal extirpation; known immunological dysfunction (human immunodeficiency virus infection); presence of ongoing infection or infective chronic diseases; severe cardiovascular disease (New York Heart Association class higher than 3) or pulmonary insufficiency (severe pulmonary emphysema, interstitial pneumonitis, arterial PO2<79 mmHg); advanced liver disease (Child-Pugh class C); synchronous or metachronous (within five years) malignancy; pregnant or lactating women; continuous systemic steroid therapy; drug addiction; previous chemotherapy, radiotherapy or immune therapy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Neutrophil activity before and after the open or laparoscopic surgery - Serum concentrations of sFas, sFasL and IL - 17. | 24 hours before surgery, 72 hours after surgery
Respiratory burst neutrophil production - Bursttest before and after open or laparoscopic surgery | 24 hours before surgery and 2 hours after surgery
Immunohistochemical detection of FasL in tumor and paratumor areas of colon cancer and normal colon mucosa taken at a distance of 10 cm from the tumor | after surgery
Immunohistochemical detection of Fas in tumor and paratumor areas of colon cancer and normal colon mucosa taken at a distance of 10 cm from the tumor | after surgery
Immunohistochemical detection of neutrophil elastase in tumor and paratumor areas of colon cancer and normal colon mucosa taken at a distance of 10 cm from the tumor | after surgery
Number of leukocytes, neutrophils, lymphocytes and neutrophils/lymphocytes ratio | 24 hours before surgery, 2 hours after surgery, 72 hours after surgery
CRP | 24 hours before surgery, 72 hours after surgery
Fe, transferrin, ferritin | 24 hours before surgery, 72 hours after surgery

SECONDARY OUTCOMES:
to determine neutrophil activity in patients with colon cancer and healthy volunteers | 24 hours before surgery, 2 hours and 72 hours after surgery
to compare the influence of laparoscopic and conventional procedures on postoperative neutrophil function | 24 hours before surgery, 2 hours and 72 hours after surgery
to determine functional activity of tumour infiltrating neutrophils | after surgery
to determine an effect of surgery on neutrophil activity | 24 hours before surgery, 2 hours and 72 hours after surgery
to determine levels sFas, sFasL and IL - 17 in serum of healthy volunteers and colon cancer patients and establish its prognostic value | 24 hours before surgery, 2 hours and 72 hours after surgery
to eludicate the relationship between serum sFas, sFasL and IL - 17 levels and clinicopathologic features of colon cancer | 24 hours before surgery, 2 hours and 72 hours after surgery
to compare the influence of laparoscopic and conventional procedures on postoperative serum sFas, sFasL and IL - 17 levels in colon cancer patients | 24 hours before surgery, 2 hours and 72 hours after surgery
to confirm the expression of FasL protein in human colorectal cancer and elucidate the relationship between FasL expression and clinicopathologic features of the disease | after surgery
to establish the prevalence of Fas in primary colon adenocarcinomas and elucidate the relationship between Fas expression and clinicopathologic features of the disease | after surgery
loss of blood during the surgery, postoperative hospital stay, morbidity, and mortality within 30 days after surgery | intraoperative and within 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Igor Stipančić, MD, PhD, Profssor, Study Chair — University Hospital Dubrava; Valentina Ratkajec, MD, Principal Investigator — University Hospital Dubrava
Locations (1):
- University Hospital "Dubrava", Zagreb, Croatia